CLINICAL TRIAL: NCT02631031
Title: A Comparative Pharmacokinetic and Pharmacodynamic Study of Morning Versus Evening Administration of Valsartan in Healthy Adults
Brief Title: Chronopharmacology of Valsartan in Normotensive Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Noha Osama Mansour, Ph.D candidate Clinical pharmacy department, Faculty of pharmacy, Ain shams University, Ain Shams University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Ph.D (No.26)
Record Dates: First submitted 2015-12-04; First posted 2015-12-15 (Estimated); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: Healthy Normotensive Volunteers
Keywords: Chronokinetics; chronodynamics; chronopharmacology; valsartan
MeSH Terms: interventions — Valsartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- morning administration (Other): administration of single oral dose valsartan (160 mg) in the morning
  Interventions: Drug: Valsartan
- evening administration (Other): administration of single oral dose valsartan (160 mg) in the evening
  Interventions: Drug: Valsartan

INTERVENTIONS:
Drug: Valsartan — single oral dose of 160 mg valsartan under fasting conditions
  Other Names: Diovan

SUMMARY:
The choice of drug administration time may affect the pharmacokinetics and/or drug response, and knowledge of any such circadian rhythm-dependent effects may help to reduce side effects or to enhance efficacy. This study designed to investigate the potential influence of the time of drug administration on the pharmacokinetics and pharmacodynamics of the valsartan in healthy subjects.

DETAILED DESCRIPTION:
International guidelines recommend the use of long acting, once-daily medications that provide 24h efficacy; they improve adherence to therapy and minimize BP variability with smoother and more consistent BP control.

Valsartan has been approved to be used once-daily, without any specification of treatment-time in package insert. Several trials have investigated the differential effects of morning versus evening administration of valsartan in hypertensive patients, however, the results of these studies were contradicting. Furthermore, the specific administration time dependent dose response curve have not been previously investigated. So, this study designed to investigate the potential influence of the time of drug administration on the pharmacokinetics and pharmacodynamics of the valsartan in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years old and not more than 45 healthy male volunteers
2. Actual weight no more than ± 30% from ideal body weight based on sex, height, and body frame
3. Who had passed all the screening parameters including physical examination, laboratory tests.
4. Who had to be able to communicate effectively with study personnel, be literate, and able to give consent.
5. diurnal active subjects with eight hour night sleep.
6. free of any drug exposure known to interfere with the pharmacokinetics/pharmacodynamics or assay of valsartan for at least 10 days prior to the study

Exclusion Criteria:

1. Treatment with any known enzyme-inducing/inhibiting agents within 30 days prior to the start of the study and throughout the study.
2. Susceptibility to allergic reactions to valsartan.
3. Any prior surgery of the gastrointestinal tract that may interfere with drug absorption.
4. Gastrointestinal diseases.
5. Renal diseases.
6. Cardiovascular diseases.
7. Pancreatic disease including diabetes.
8. Hepatic diseases.
9. Hematological disease or pulmonary disease
10. Abnormal laboratory values.
11. Subjects who have donated blood or who have been involved in multiple dosing study requiring a large volume of blood (more than 500 ml) to be drawn within 6 weeks preceding the start of the study.
12. Nocturnal active subjects

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-11; Primary Completion 2016-10 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters | blood samples will be collected for 48 hour after drug administration
  Maximum plasma concentration (Cmax),
Pharmacokinetic parameters | blood samples will be collected for 48 hour after drug administration
  Area under the curve (AUC).
Pharmacokinetic parameters | blood samples will be collected for 48 hour after drug administration
  elimination half life (T1/2)
pharmacodynamic parameter | Blood samples will be measured at prespecified time points for 48 hour after drug administration
  systolic blood pressure (mm Hg) ,diastolic blood pressure (mm Hg)
pharmacodynamic parameter | Blood samples will be measured at prespecified time points for 48 hour after drug administration
  Heart rate (beat/min)

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No